CLINICAL TRIAL: NCT00000523
Title: Optimal Exercise Regimens for Persons at Increased Risk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 42
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-01

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia | interventions — Exercise

INTERVENTIONS:
Behavioral: exercise

SUMMARY:
To assess exercise training adherence and compliance over two years in subjects who were at relatively high risk for coronary artery disease. Also, to test strategies for improving adherence and compliance and to assess the effect of exercise training.

DETAILED DESCRIPTION:
BACKGROUND:

Regular physical exercise is associated with lower coronary heart disease mortality, favorably affects coronary risk factors, and increases cardiovascular functional capacity. Fewer than one-third of Americans engage in regular physical exercise and only 20 percent of men and 10 percent of women over age 45 do so. This is largely because effective strategies for increasing the exercise habit in a broadly-based segment of Americans have not been developed. This study applied physiological and behavioral knowledge derived in numerous laboratories over the past 10-15 years to a clinical setting.

DESIGN NARRATIVE:

Following stratification by gender and cigarette smoking status, subjects were randomized to one of four groups: home exercise of moderate intensity which was individually monitored; home exercise of high intensity which was individually monitored; exercise of high intensity which was group supervised; and a no program control group. The intervention program was conducted for one year followed by a one-year maintenance program. Main outcome measures included treadmill exercise test performance, exercise participation rates, and heart disease risk factors. Variables measured over two years included plasma lipids, lipoproteins, apoproteins, lipase activity, glucose and insulin, sex hormones, cardiovascular reactivity to psychological stress, cigarette smoking, nutrient intake, psychological status, and cardiovascular functional capacity.

ELIGIBILITY:
Sedentary men and women, ages 50 to 65. Women were postmenopausal and not taking hormone replacement therapy. All subjects were free from, but at increased risk for, coronary heart disease.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1986-04

REFERENCES:
- [Background] King AC, Haskell WL, Taylor CB, Kraemer HC, DeBusk RF. Group- vs home-based exercise training in healthy older men and women. A community-based clinical trial. JAMA. 1991 Sep 18;266(11):1535-42. PMID 1880885